CLINICAL TRIAL: NCT02384993
Title: Aerobic Exercise for Alzheimer's Disease Prevention in At-Risk Middle-Aged Adults
Brief Title: aeRobic Exercise and Cognitive Health
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1434; 2014-NIRGD-305257 (Other Grant/Funding Number: Alzheimer's Association); A534255 (Other: UW Madison); SMPH\MEDICINE\GER-AD DEV (Other: UW Madison)
Record Dates: First submitted 2015-02-25; First posted 2015-03-10 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Disease; Aging
Keywords: Alzheimer's Disease; Dementia; aerobic exercise; physical activity; exercise; neuroimaging
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Physical Activity (Experimental): Those assigned to the enhanced physical activity group will train 3-4 days per week with the goal of attaining current public health recommendations of 150 minutes of moderate intensity exercise by the 7th week of training, and maintaining this level of exercise for the remainder of the 26-week intervention. A gradual increase in exercise intensity and duration will be used throughout this twenty-six week exercise intervention, with the initial speed and duration calibrated to each participant's baseline aerobic capacity. Training will occur in individual sessions supervised by exercise specialists with the appropriate education and experience. Each training session will begin with an appropriate warm-up, slowly build up, and end with an appropriate cool down period.
  Interventions: Behavioral: Enhanced Physical Activity
- Usual Physical Activity (No Intervention): All study participants randomized to the usual physical activity group will receive education from study staff about the importance of maintaining a healthy and active lifestyle. They will receive standardized literature such as "Exercise & Physical Activity: Your Everyday Guide from the National Institute on Aging". These booklets provide vetted and reliable information for older adults on how to exercise. Participants assigned to the usual physical activity group will not be provided additional support or guidance with an exercise program.

INTERVENTIONS:
Behavioral: Enhanced Physical Activity — This is a 26-week aerobic exercise intervention. The primary mode of training is treadmill walking, with the initial speed and duration calibrated to each participant's baseline aerobic capacity. Participants will train 3-4 days per week with the goal of attaining 150+ minutes of exercise per week by the seventh week. Exercise will be set between 50-60% of maximum heart rate reserve for weeks 1-4, 60-70% for weeks 5-8, and 70-80% for weeks 9-26. Exercise duration will be approximately 15-20 minutes per session during the first week and then increase by 5 minutes each week until a duration of approximately 38-50 minutes per session is reached. Each training session will begin with a 5-minute warm-up and end with a 5-minute recovery period.
  Other Names: Aerobic Exercise (EXER)
  Arms: Enhanced Physical Activity

SUMMARY:
The purpose of the aeRobic Exercise and Cognitive Health (REACH) study is to understand how an aerobic exercise intervention might help promote brain health and cognition, thereby delaying the onset of clinical symptoms of Alzheimer's disease.

DETAILED DESCRIPTION:
The prevalence and costs associated with Alzheimer's disease (AD) are projected to increase exponentially owing to the unprecedented expansion in the elderly segment of the United States' population. Given this looming specter, delaying the onset of AD symptoms and curbing the progression of the underlying disease process has become a national public health imperative. Delaying symptom onset by as little as 5 years could reduce the prevalence of AD by half. Unfortunately, currently available drug treatments for AD are not curative. Similarly, clinical trials testing novel disease-modifying therapeutics have been disappointing. The urgency of alternative approaches for halting the global crisis posed by AD cannot be overstated.

Animal studies have demonstrated that aerobic exercise (EXER) is a low-cost, low-risk intervention capable of altering the AD pathological process. Randomized controlled trials (RCTs) of EXER in older adults have also revealed its beneficial effects on AD-relevant measures such as brain glucose metabolism and memory/executive function. Importantly, a recent evidence review found that of 7 key modifiable risk factors for AD, physical activity had the highest impact on reducing the national prevalence of AD. However, there are presently no RCTs examining the effects of EXER in middle-aged, asymptomatic individuals at increased risk of AD. This is an important knowledge gap for several reasons. Interventions to halt the AD pathological cascade are more likely to be effective if implemented prior to pervasive neuronal damage. Secondly, persons with specific risk factors for developing AD (such as parental family history (FH)) represent a choice target population for any credible attempts at reducing the growing burden of AD. Lastly, a key limitation of prior EXER RCTs is the failure to adequately account for participants' physical activity levels outside of the intervention.

Accordingly, the main objective of this study is to pilot a 26-week trial of EXER among asymptomatic, middle-aged adults with and without family history (FH) of AD enrolled in the Wisconsin Registry for Alzheimer's Prevention (WRAP) or the Wisconsin Alzheimer's Disease Research Center (WADRC). The investigators' near-term goal is to assess the feasibility and acceptability of this structured intervention and preliminarily evaluate (i) its effect on AD-relevant outcomes such as glucose metabolism and (ii) the mechanism for such effects. The investigators' longer-term goal is to use the data gathered via this pilot to further refine the intervention, estimate effect sizes for key outcomes, and seek NIH funding for a longer and more definitive assessment of whether EXER can effectively curtail AD progression in midlife. The specific aims are:

AIM 1: Determine the feasibility and acceptability of a 26-week, 3-4 days per week, structured EXER regimen among middle-aged adults with FH of AD. Hypothesis: The investigators will successfully enroll the 30 participants (15 each in EXER and usual physical activity groups) targeted for this study. At least 90% of the participants within the EXER group, called the enhanced physical activity group, will complete ≥80% of scheduled training sessions.

AIM 2: Preliminarily characterize the effect of the EXER intervention on AD-related brain alteration. Hypothesis: Compared to participants randomized to the usual physical activity group, those randomized to the enhanced physical activity group will demonstrate preserved brain glucose metabolism. Similar effects will be seen in secondary outcomes including cerebral blood flow, hippocampal volume, vascular health, memory/executive function, and mood.

AIM 3: Preliminarily evaluate (i) the biological mechanisms by which EXER affects brain health and cognition, and (ii) the individual difference factors that potentially moderate EXER's effects. Hypotheses: (i) Persons in the enhanced physical activity group will exhibit significant increases in circulating neurotrophins and improved cardiorespiratory fitness, and (ii) the beneficial effects of EXER will be more pronounced for participants with decreased sedentary behaviors outside of the intervention (measured via accelerometry).

AIM 4: Preliminarily determine whether EXER improves vascular health. Hypothesis: Individuals in the enhanced physical activity group will exhibit comparatively increased cerebral blood flow, and improved endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 at baseline visit.
* Must be currently physically inactive (i.e. not meeting national guidelines of 150+ minutes per week of moderate exercise).
* Participant is not pregnant at the time of the positron emission tomography (PET) and magnetic resonance (MR) imaging exams.
* Willing and able to complete all assessments and exercise intervention faithfully.
* Fluent and proficient in English language and capable of completing neuropsychological testing in English.
* Participant must have physician clearance to participate in this study.

Exclusion Criteria:

* Any significant neurologic disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma (10 min or more of loss of consciousness) followed by persistent neurologic deficits or known structural brain abnormalities.
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, body. X-ray may be used to establish suitability for MRI.
* Inability to complete exercise test due to medical restrictions such as hip surgery, knee surgery, arthritis, or other orthopedic concerns that prevent being able to walk on a treadmill, type I or II diabetes mellitus, and documented vascular disease such as coronary artery disease.
* Clinically significant findings from the exercise test that prohibit participation in moderate intensity exercise (i.e. 3rd degree heart block).
* Current Axis I DSM-IV disorder including but not limited to major depression within the past two years, history of bipolar I disorder, history of schizophrenia spectrum disorders (DSM IV criteria).
* History of alcohol or substance abuse or dependence (DSM IV criteria).
* Any significant systemic illness or unstable medical condition that could affect cognition, CBF or BOLD, or cause difficulty complying with the exam. History of chemotherapy, thyroid disease, or renal insufficiency are excluded.
* Severe untreated hypertension (>200/100mmHG).
* Participants who do not have the cognitive competence and legal capacity to make informed medical decisions are excluded at entry. If a participant experiences significant cognitive decline during the study such that they no longer have medical decision making capacity the investigators will enact procedures that have been approved locally by the IRB and legal counsel at the University of Wisconsin-Madison: A) use their initial expressed and written consent as an indicator of willingness to continue to participate in the study; AND B) require that they provide assent at the time of follow-up visits witnessed and counter signed by their caregiver; AND C) signed consent from the patient's legally authorized representative.
* Current use of antipsychotic medications such as non-SSRI antidepressants, neuroleptics, chronic anxiolytics, or sedative hypnotics, as well as some cardiac glycosides such as Digoxin.
* Investigational agents are prohibited.
* Exceptions to these criteria will be rare but may be considered on a case-by-case basis at the discretion of the investigators in consultation with study physicians.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozioma C. Okonkwo, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health & Human Services. National Plan to Address Alzheimer's Disease: 2014 Update. Available at http://aspe.hhs.gov/daltcp/napa/NatlPlan2014.pdf. Accessed February 17, 2015.
- [Background] Khachaturian ZS, Khachaturian AS. Prevent Alzheimer's disease by 2020: a national strategic goal. Alzheimers Dement. 2009 Mar;5(2):81-4. doi: 10.1016/j.jalz.2009.01.022. No abstract available. PMID 19328433
- [Background] Sperling RA, Jack CR Jr, Aisen PS. Testing the right target and right drug at the right stage. Sci Transl Med. 2011 Nov 30;3(111):111cm33. doi: 10.1126/scitranslmed.3002609. PMID 22133718
- [Background] Adlard PA, Perreau VM, Pop V, Cotman CW. Voluntary exercise decreases amyloid load in a transgenic model of Alzheimer's disease. J Neurosci. 2005 Apr 27;25(17):4217-21. doi: 10.1523/JNEUROSCI.0496-05.2005. PMID 15858047
- [Background] Wu CW, Chang YT, Yu L, Chen HI, Jen CJ, Wu SY, Lo CP, Kuo YM. Exercise enhances the proliferation of neural stem cells and neurite growth and survival of neuronal progenitor cells in dentate gyrus of middle-aged mice. J Appl Physiol (1985). 2008 Nov;105(5):1585-94. doi: 10.1152/japplphysiol.90775.2008. Epub 2008 Sep 18. PMID 18801961
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Plymate SR, Fishel MA, Watson GS, Cholerton BA, Duncan GE, Mehta PD, Craft S. Effects of aerobic exercise on mild cognitive impairment: a controlled trial. Arch Neurol. 2010 Jan;67(1):71-9. doi: 10.1001/archneurol.2009.307. PMID 20065132
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Jarvik L, LaRue A, Blacker D, Gatz M, Kawas C, McArdle JJ, Morris JC, Mortimer JA, Ringman JM, Ercoli L, Freimer N, Gokhman I, Manly JJ, Plassman BL, Rasgon N, Roberts JS, Sunderland T, Swan GE, Wolf PA, Zonderman AB. Children of persons with Alzheimer disease: what does the future hold? Alzheimer Dis Assoc Disord. 2008 Jan-Mar;22(1):6-20. doi: 10.1097/WAD.0b013e31816653ac. PMID 18317242
- [Result] Gaitan JM, Boots EA, Dougherty RJ, Oh JM, Ma Y, Edwards DF, Christian BT, Cook DB, Okonkwo OC. Brain Glucose Metabolism, Cognition, and Cardiorespiratory Fitness Following Exercise Training in Adults at Risk for Alzheimer's Disease. Brain Plast. 2019 Dec 26;5(1):83-95. doi: 10.3233/BPL-190093. PMID 31970062
- See also: U.S. Department of Health & Human Services. National Plan to Address Alzheimer's Disease: 2014 Update — https://aspe.hhs.gov/sites/default/files/private/pdf/102496/NatlPlan2014%20with%20Note.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Physical Activity: Usual Physical Activity: Participants in this group will receive education from study staff about the importance of maintaining a healthy and active lifestyle. They will receive standardized literature such as "Exercise & Physical Activity: Your Everyday Guide from the National Institute on Aging". These booklets provide vetted and reliable information for older adults on how to exercise. Participants assigned to the usual physical activity group will not be provided additional support or guidance with an exercise program.
- Enhanced Physical Activity: Enhanced Physical Activity: Participants in this group will engage in a 26-week treadmill walking aerobic exercise intervention. The initial speed and duration will be calibrated to each participant's baseline aerobic capacity. Participants will train 3-4 days per week with the goal of attaining current public health recommendations of 150 minutes of moderate intensity exercise by the 7th week of training and maintaining this level of exercise for the remainder of the 26-week intervention. Exercise will be set at 50-60% of maximum heart rate reserve for weeks 1-4, 60-70% for weeks 5-8, and 70-80% for weeks 9-26. Exercise duration will be 15-20 minutes per session during the first week and then increase by 5 minutes each week until a duration of approximately 38-50 minutes per session is reached. Each training session will begin with a 5-minute warm-up and end with a 5-minute recovery period. Training will occur in individual sessions supervised by exercise specialists.
Period: Overall Study
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Measures reported for participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Physical Activity | Enhanced Physical Activity | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Count of Participants; unit: Participants]
  Age: 50-59 years | 4 | 1 | 5
  Age: 60-69 years | 7 | 9 | 16
  Age: 70-79 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years of Education [Mean (Standard Deviation); unit: years] | 16.67 (2.57) | 16.58 (2.47) | 16.62 (2.46)
Number of Participants with APOE e4 positive [Count of Participants; unit: Participants] — Apolipoprotein E (APOE) is a protein in the body used to metabolize fat, the presence of the epsilon 4 allele (APOE e4)is correlated to increased Alzheimer's and cardiovascular disease risk.
  Participants | 5 | 4 | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI)
  kg/m^2 | 29.38 (5.96) | 29.37 (4.93) | 29.37 (5.35)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 128.50 (19.65) | 121.88 (18.39) | 125.19 (18.92)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 79.92 (9.47) | 75.33 (10.20) | 77.63 (9.90)
Number of Participants with Parental History of Alzheimer's Disease [Count of Participants; unit: Participants] | 12 | 12 | 24
MMSE [Mean (Standard Deviation); unit: scores on a scale] — Mini-Mental State Examination (MMSE) is a question scored from 0-30 where scores of 0-17 indicate severe cognitive impairment, 18-23 indicate mild cognitive impairment, and 24-30 indicate no cognitive impairment.
  scores on a scale | 29.67 (0.49) | 29.58 (0.67) | 29.62 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: Percentage of Sessions Completed by Enhanced Physical Activity Group
Description: This intervention will be considered acceptable if participants who complete the Enhanced Physical Activity intervention, complete ≥80% of scheduled training sessions.
Time Frame: up to 26 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Sessions
Arm/Group | Enhanced Physical Activity
Number analyzed (Participants) | 11
Percentage of Sessions | 99.2 (2.7)

2. Primary Outcome: Feasibility: Percentage of Participants Who Completed the Study
Description: Feasibility is in part defined as at least 90% of enrolled participants completed the study.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 12
Participants | 12 | 11

3. Primary Outcome: Cerebral Glucose Metabolism as Measured by FDG PET Scanning
Description: Changes in cerebral glucose metabolism will be assessed using fluorodeoxyglucose (FDG) positron emission tomography (PET) scanning. This method measures the brain's use of blood sugar while in a resting state. Measurements were taken in the posterior cingulate cortex (PCC). An increase in this measure indicates an increase in the brain's uptake and usage of blood sugar.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
arbitrary units
  baseline | 1.49 (0.04) | 1.50 (0.03)
  26 weeks | 1.52 (0.04) | 1.54 (0.04)

4. Secondary Outcome: Ultrasound-Measured Cerebral Blood Flow - Mean Flow Velocity
Description: Cerebral blood flow velocity changes in the middle cerebral artery will be measured using Transcranial Doppler ultrasound imaging.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Median (Inter-Quartile Range); unit: cm/second
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 11 | 9
cm/second
  Baseline | 45.05 [42.59 to 47.51] | 41.13 [33.97 to 48.29]
  26 Weeks | 49.47 [42.16 to 56.78] | 45.85 [37.35 to 54.36]

5. Secondary Outcome: California Verbal Learning Test-II Total Score
Description: The California Verbal Learning Test-II assesses cognitive function. Higher scores indicate more words recalled. Scores range from 0 to 100.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
words
  baseline | 49.58 (11.06) | 53.18 (7.99)
  26 weeks | 53.33 (9.18) | 60.64 (9.04)

6. Secondary Outcome: Delis-Kaplan Executive Function System Color Word Interference (D-KEFS CWI) Score
Description: The D-KEFS CWI will be used to measure executive function. Lower times indicate improved executive function. Scores range from 0 to 90.
Time Frame: up to 26 weeks (measured at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
seconds
  baseline | 60.00 (11.71) | 64.82 (15.11)
  26 weeks | 60.00 (11.99) | 57.64 (11.96)

7. Secondary Outcome: Mini Mental State Examination (MMSE) Score
Description: The Mini Mental State Examination (MMSE) measures global cognitive function. Scores range from 0 to 30. Higher scores indicate better cognitive function.
Time Frame: up to 26 weeks (assessed at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
scores on a scale
  baseline | 29.67 (0.49) | 29.55 (0.69)
  26 weeks | 29.08 (1.24) | 29.55 (0.52)

8. Secondary Outcome: California Verbal Learning Test-II Long Delay Score
Description: The California Verbal Learning Test-II assesses cognitive function. Long delay is a test where there is a 20 minute time period between initial word list presented and recall. Higher scores indicate more words recalled. Scores range from 0 to 20.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
words
  baseline | 10.83 (2.83) | 12.00 (2.72)
  26 weeks | 11.42 (3.26) | 14.00 (1.73)

9. Secondary Outcome: Profile of Mood States (POMS) Score
Description: The Profile of Mood States was used to assess mood. POMS is divided into six subscales including tension-anxiety (9 items, score range: 0-36), depression (15 items, range: 0-60), anger-hostility (12 items, range: 0-48), vigor-activity (8 items, range: 0-32), fatigue (7 items, range: 0-28), and confusion-bewilderment (7 items, range: 0-28). Total mood disturbance is calculated by adding five of the six subscales (Tension, Depression, Anger, Fatigue, and Confusion) and subtracting Vigor (Scores range from -32 to 200). Lower scores typically indicate more steady mood profiles. Higher scores indicate more mood disturbance.
Time Frame: up to 26 weeks (assessed at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
score on a scale
  Baseline Tension | 8.00 (2.92) | 7.67 (3.11)
  Post-intervention Tension | 8.64 (3.41) | 6.00 (3.82)
  Baseline Depression | 5.17 (6.60) | 4.83 (6.64)
  Post-intervention Depression | 5.36 (5.52) | 3.27 (5.53)
  Baseline Anger | 3.17 (4.49) | 5.50 (4.98)
  Post-intervention Anger | 4.27 (3.41) | 3.82 (5.10)
  Baseline Vigor | 16.83 (6.31) | 16.25 (6.86)
  Post-intervention Vigor | 16.25 (6.86) | 15.36 (4.74)
  Baseline Fatigue | 4.92 (3.55) | 6.58 (5.25)
  Post-intervention Fatigue | 7.64 (4.15) | 5.91 (4.70)
  Baseline Confusion | 5.17 (2.95) | 6.83 (2.52)
  Post-intervention Confusion | 5.55 (3.05) | 5.45 (3.17)
  Baseline Total Mood Disturbance | 9.58 (19.71) | 15.17 (19.94)
  Post-intervention Total Mood Disturbance | 16.09 (15.64) | 7.55 (20.47)

10. Secondary Outcome: Change in Hippocampal Volume
Description: Hippocampal volume will be assessed using T1-weighted 3T MRI images.
Time Frame: up to 26 weeks (assessed at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: mm cubed
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
mm cubed | -23.67 (222.50) | -33.64 (177.00)

11. Other Pre Specified Outcome: Ancillary Neuroimaging Measures
Description: Ancillary neuroimaging measures include MRI brain scans of blood flow and brain structure.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Cardiorespiratory Fitness Measured by Peak Oxygen Consumption (VO2peak)
Description: The investigators will examine Cardiorespiratory Fitness by measuring VO2peak on a graded treadmill test - after participants fasted for 12-hours.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Mean (Standard Error); unit: mL/kg/min
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
mL/kg/min
  baseline | 25.74 (6.58) | 23.57 (4.97)
  26 weeks | 27.18 (6.05) | 27.46 (4.71)

13. Other Pre Specified Outcome: Brain Derived Neurotrophic Factor
Description: The investigators will examine levels of Brain Derived Neurotrophic Factor to assess changes in blood neurotrophic levels.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Vascular Endothelial Growth Factor
Description: Levels of Vascular Endothelial Growth Factor will be assessed to identify changes in vascular health.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Arterial Plaque Presence
Description: Changes in plaque presence will be measured using Comprehensive Carotid Ultrasound.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Subclinical Atherosclerosis Burden
Description: Changes in subclinical atherosclerosis burden will be measured using Carotid Intima-Media Thickness Ultrasound.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Endothelial Function
Description: Endothelial function changes will be assessed via ultrasound using Brachial Artery Reactivity Testing.
Time Frame: over 26 weeks (assessed at baseline visit and at week-26 visit)
Measure: Mean (Standard Deviation); unit: Percentage of dilation
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 9
Percentage of dilation
  Baseline | 2.22 (1.78) | 1.86 (0.93)
  26 Weeks | 2.71 (1.69) | 2.33 (1.71)

18. Other Pre Specified Outcome: Sedentary Behavior Measured Via Accelerometer
Description: Participants wore a triaxial accelerometer (GT3X+, Actigraph LLC, Pensacola, FL) for seven consecutive days to record free-living PA and sedentary behavior before and after the intervention.
Time Frame: up to 26 weeks (measured at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: minute/day
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
minute/day
  Baseline | 670.73 (27.2) | 726.0 (22.9)
  26 weeks | 690.1 (26.7) | 698.6 (27.1)

19. Other Pre Specified Outcome: Moderate to Vigorous Physical Activity (MVPA)
Description: Participants wore a triaxial accelerometer (GT3X+, Actigraph LLC, Pensacola, FL) for seven consecutive days to record free-living physical activity before and after the intervention.
Time Frame: up to 26 weeks (assessed at baseline and 26 weeks)
Measure: Mean (Standard Deviation); unit: minute/day
Arm/Group | Usual Physical Activity | Enhanced Physical Activity
Number analyzed (Participants) | 12 | 11
minute/day
  baseline | 78.97 (10.19) | 60.58 (7.08)
  26 weeks | 69.3 (8.37) | 89.05 (15.48)

ADVERSE EVENTS:
Time Frame: up to 26 weeks
Arm/Group | Enhanced Physical Activity | Usual Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Physical Activity (N=12) | Usual Physical Activity (N=12)
Hip Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes